CLINICAL TRIAL: NCT06009952
Title: EFFECT OF CYOLIPOLYSIS DEVICE WITH VEGAN DIET VERSUS CAVITATION DEVICE WITH VEGAN DIET ON SERUM LIPID PROFILE IN WOMEN WITH CENTRAL OBESITY
Brief Title: EFFECT OF CYOLIPOLYSIS VERSUS CAVITATION WITH VEGAN DIET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Abdelwhab, EFFECT OF CYOLIPOLYSIS DEVICE WITH VEGAN DIET VERSUS CAVITATION DEVICE WITH VEGAN DIET ON SERUM LIPID PROFILE IN WOMEN WITH CENTRAL OBESITY, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004629
Record Dates: First submitted 2023-08-20; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Healthy Adult Women
MeSH Terms: interventions — Diet, Vegan

STUDY DESIGN:
Intervention Model Description: •Pre/ posttest randomized controlled trial design.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): •Group A will receive cryolipolysis with vegan diet,
  Interventions: Other: Cryolipolysis and cavitation devices with vegan diet
- Group B (Experimental): Group B will receive cavitation with vegan diet
  Interventions: Other: Cryolipolysis and cavitation devices with vegan diet
- Group C (Experimental): Group C will receive vegan diet only.
  Interventions: Other: Cryolipolysis and cavitation devices with vegan diet

INTERVENTIONS:
Other: Cryolipolysis and cavitation devices with vegan diet — Cryolipolysis: In all cases of group A, (OPTIMIZED CRYOLIPOLYSIS 360 DEVICE, model: AF2000-02, made in china) uses a vacuum-based huge applicator (Cool Max) and vacuum medium applicators (either CoolCore or Cool- Curveþ) for the abdomen (30 minutes session twice monthly for three successive3 months).
  •Cavitation: in all cases of group B, (CAVITATION DEVICE, Item No.:AU61, Made in china) of 45 KHz frequency (30 min twice weekly for three successive3 months).

SUMMARY:
Pre/ posttest randomized controlled trial design.

In this study all females will be randomly assigned into three groups (20 for each group).

* Group A will receive cryolipolysis with vegan diet,
* Group B will receive cavitation with vegan diet and
* Group C will receive vegan diet only.

DETAILED DESCRIPTION:
Treatment Protocol:

1. Cryolipolysis: In all cases of group A, (OPTIMIZED 360 CRYOLIPOLYSIS DEVICE, model: AF2000-02, made in china) uses a vacuum-based huge applicator (Cool Max) and vacuum medium applicators (either CoolCore or Cool- Curveþ) for the abdomen (30 minutes session twice monthly for three successive3 months). The subcutaneous-fat layer in the regions of the abdomen will be treated with cryolipolysis. It will be cooled to (-8∘ C) for 30 minutes with the cryolipolysis device Areas will be treated with either the medium or large applicator, based on the size of the localized fat area and the anatomical limitations of the applicator placement.

The treatment sessions will be performed with the subjects comfortably positioned in the dorsal decubitus position with a 45∘ stretcher inclination or in the lateral decubitus position. The curved vacuum applicator will be positioned in the center of the treatment area, and vacuum suction will be initiated. The vacuum itself will be fixed the applicator over the treatment area, and pillows will be supported the applicator during the entire treatment.

The cavitation instrument generates low-frequency ultrasonic pulsed waves 45kHz through a transducer with a diameter of 45 mm and a power of 3 watts/cm2. The individual will be positioned in a comfortable supine posture, and the transducer will be placed on an abdominal region already coated with conduction gel. For three months, abdomen area will be treated with one 30-minute session twice weekly. The patient will be treated in a relaxed supine resting position.

Diet intervention:

A well-balanced vegan diet( Lacto-ovo vegetarian diet) excludes meat, fish and poultry, but allows dairy products and eggs.Vegetarian diet: Daily amounts will be based on 2,000-calorie diet.

It should be characterized by a high intake of fiber (≥45-60 g/day), a moderate intake of protein (<15% of energy), and a low intake of total fat (10-20% of energy), saturated fat (≤5% of energy), free sugars (<5% of energy) and sodium (1500 mg/day). The required supplementation must include reliable sources of vitamin B12 for the whole year and vitamin D in the winter months (vitamin fortified foods and/or a supplement), and optionally may include EPA/DHA throughout the year.

ELIGIBILITY:
Inclusion Criteria:

* 1-Their ages will be ranged between 25-40 year old.

  2-Their body mass index will be ranged between 35:39.9 kg/m2. 3-All women will have central obesity in abdominal region their waist circumference >102cm (40in).

  4-The average number of previous deliveries for all women is 4 times. 5-Included fasting serum lipid profile will be in borderline and high risk ranges.

Exclusion Criteria:

* Epileptic fits.

  * Cardiac affection and using pace maker.
  * Heavy Smokers.
  * Renal, liver or endocrinal disorder.
  * Pulmonary or lung diseases.
  * Pregnant women.
  * Patients receiving any drug therapy such as lipid lowering therapy, vitamins and antioxidants.
  * Weight reduction medications

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-31 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Fasting serum lipid profile | Three months
  Pre/post Fasting serum lipid profile

SECONDARY OUTCOMES:
Waist circumference | Three months
  All women will have central obesity in abdominal region their waist circumference >102cm (40in).

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: One year after completion the study
Access Criteria: Students and scientific researchers will be allowed to access